CLINICAL TRIAL: NCT07313761
Title: A Phase 1, Open-label, Randomized, Parallel Group Study to Assess the Relative Bioavailability of Maridebart Cafraglutide (AMG 133) as Two Subcutaneous Presentations in Participants Living With Overweight or Obesity
Brief Title: A Trial to Compare the Extent to Which Maridebart Cafraglutide (AMG 133) is Made Available in the Body When Administered Using Two Subcutaneous Presentations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210268
Record Dates: First submitted 2025-12-19; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Overweight; AMG 133; Maridebart cafraglutide; MariTide
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide SC Presentation 1 (Experimental): Participants will receive a single dose of maridebart cafraglutide administered using SC presentation 1.
  Interventions: Drug: Maridebart Cafraglutide
- Maridebart Cafraglutide SC Presentation 2 (Active Comparator): Participants will receive a single dose of maridebart cafraglutide administered using SC presentation 2.
  Interventions: Drug: Maridebart Cafraglutide

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133

SUMMARY:
The main objective of this trial is to evaluate the pharmacokinetics (PK) of maridebart cafraglutide administered as a single dose using two different SC presentations in participants living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, between 18 and 60 years of age, inclusive.

   a. Females must not be pregnant or lactating.
2. Body mass index between 25.0 and <40.0 kg/m^2.
3. Have a stable body weight (<5 kg self-reported change) within 3 months before screening, as assessed by the investigator (or designee) based on participant self-report.

Exclusion Criteria:

1. History or evidence, at screening or check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the investigator (or designee), would pose a risk to participant safety or interfere with the trial evaluation, procedures, or completion. Participants with clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) as assessed by the investigator (or designee) will be excluded.
2. History of or active diabetes (regardless of type, with the exception of a history of gestational diabetes) or hemoglobin A1C ≥6.5% (≥48 mmol/mol).
3. History or evidence of endocrine disorder (eg, Cushing's Syndrome) that can cause obesity.
4. History of acute or chronic pancreatitis within 1 year prior to check-in, or elevation in serum lipase/amylase (>2 x the upper limit of normal) at screening or a fasting serum triglyceride level of >500 mg/dL at screening.
5. Malignancy, except nonmelanoma skin cancers or cervical or breast ductal carcinoma in situ, within the last 5 years.
6. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
7. History or current signs or symptoms of cardiovascular disease (aside from controlled hypertension and controlled dyslipidemia), including but not limited to myocardial infarction, congenital heart disease, valvular heart disease, coronary revascularization, or angina.
8. History or evidence of clinically significant arrhythmia at screening, including any clinically significant findings on the ECG taken at screening or check-in.
9. History of hypersensitivity, intolerance, or allergy to AMG 133 or related/similar compounds or their ingredients.
10. Estimated glomerular filtration rate ≤60 mL/min/1.73 m^2, as calculated by the Chronic Kidney Disease Epidemiology (CKD EPI) equation at screening or check-in.
11. Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before check-in.
12. Current use or prior use of any glucagon-like peptide-1 receptor (GLP-1R) agonist, or gastric inhibitory polypeptide receptor (GIPR) agonist or antagonist within the past 3 months prior to check-in.
13. Current or prior use of all herbal medicines (eg, St. John's wort), vitamins, and supplements consumed by the participant within the 30 days prior to enrollment, unless deemed acceptable by the investigator (or designee) and in consultation with the medical monitor, as appropriate.
14. Participant has received a dose of an investigational drug within the past 30 days or 5 half-lives, whichever is longer, prior to check-in.
15. Have previously completed or withdrawn from this trial or any other trial investigating AMG 133 or have previously received the investigational product.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Infinity (AUCinf) of AMG 133 | Up to Day 120
AUC From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of AMG 133 | Up to Day 120
Maximum Observed Plasma Concentration (Cmax) of AMG 133 | Up to Day 120

SECONDARY OUTCOMES:
Number of Participants who Experienced Treatment-emergent Adverse Events (TEAEs) | Day 1 to Day 120
Number of Participants who Experienced Serious AEs (SAEs) | Screening to Day 120 (up to 148 days)
Number of Participants with Positive Anti-AMG 133 Antibodies | Up to Day 120

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - CenExel Collaborative Neuroscience Research, LLC Los Alamitos, Los Alamitos, California
  - Clinical Pharmacology Of Miami, LLC, Miami, Florida
  - Ohio Clinical Trials, Inc., Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com